CLINICAL TRIAL: NCT06622044
Title: Accommodation and Vergence Exercises Versus Prism Treatment for Small-angle Acute Acquired Concomitant Esotropia
Brief Title: Vision Therapy Versus Prism Treatment in Small-angle Acute Acquired Concomitant Esotropia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-ATAACE
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Esotropia
Keywords: Vision Therapy; Acute Acquired Concomitant Esotropia
MeSH Terms: conditions — Esotropia | interventions — PRDM6, protein, mouse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vision therapy group (Experimental): Accommodation facility exercises and divergence exercises
  Interventions: Other: Vision therapy group
- Prism group (Active Comparator): wearing prism glasses
  Interventions: Other: Prism

INTERVENTIONS:
Other: Vision therapy group — accommodation and vergence exercise
  Arms: Vision therapy group
Other: Prism — wearing prism glasses
  Arms: Prism group

SUMMARY:
This is a single-center, randomized controlled clinical trial to compare the effectiveness of vision therapy and prism wearing for the treatment of small-angle acute acquired concomitant esotropia.

DETAILED DESCRIPTION:
Acute acquired concomitant esotropia (AACE) belongs to the category of concomitant strabismus. It is characterized by sudden onset, often accompanied by diplopia, and no change in the strabismus angle of each eye position. In recent years, with the increase in the use of smartphones and other screen devices, the incidence of AACE has been on the rise. Commonly used treatments in clinical practice include surgical treatment, botulinum toxin injection into the medial rectus muscle, and prism treatment. Patients with large-angle esotropia generally require surgical intervention to fundamentally correct patients eye positions and eliminate diplopia. However, surgical treatment requires waiting for six months in order to performed after the strabismus degree is stable. There are also risks of intraoperative trauma and secondary surgery. Patients with early and small-angle esotropia often choose prism treatment.

The principle of prism treatment is light refraction. After light is refracted through a prism, it falls on the fovea of the strabismic eye, eliminating diplopia. In the treatment of AACE, the main target population of prisms is patients with mild strabismus (the strabismus angle is usually less than 25 PD). Wearing prisms can eliminate diplopia and relieve related symptoms, but it does not really correct the strabismus problem.

The high incidence of AACE is related to excessive close work and use of electronic products. Excessive close eye use can lead to accommodative dysfunction. Studies have found that AACE patients have abnormal accommodative function. The accommodative function of AACE patients is weaker than normal, and the accommodation convergence to accommodation (AC/A) ratio is higher than normal. During clinical diagnosis and treatment, the accommodative function of AACE patients was examined and it was found that there was indeed abnormal accommodative function. Based on scientific research findings and the actual basis of clinical practice, improving accommodative function through accommodative training may be a good treatment option for early and small-angle AACE patients. However, existing studies have not fully explored the effectiveness and safety of accommodative exercise in the treatment of small-angle AACE, and there has been no study comparing the therapeutic outcomes of accommodative training and prism treatment on small-angle AACE.

In order to better guide clinical practice, we conducted a randomized controlled study to objectively evaluate and compare the therapeutic effects of accommodative training and prism therapy on AACE. It is expected that the research results will provide more treatment options for AACE patients and provide important guidance for clinical selection of appropriate methods to treat small-angle AACE.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 10-40 years (including 10 years and 40 years);
2. Best-corrected visual acuity no worse than 20/20 for both eyes;
3. Deviation angle less than 15 prism diopters (including 15 prism diopters);

Exclusion Criteria:

1. Organic eye diseases;
2. Lesions of the brain;
3. Receiving esotropia therapy(including surgery and prism treatment)
4. Devation angle reducing more than 10 prism diopters after refractive correction

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Change in deviation angle at distance and near | 1 weeks, 4weeks, 12 weeks, 24 weeks
  the deviation angle measured using the alternate prism cover test

SECONDARY OUTCOMES:
Changes in stereopsis | 1 weeks, 4weeks, 12 weeks, 24 weeks
  Near and far stereopsis measured with Randot Stereotest pattern
Changes in accommodation facility | 1 weeks, 4weeks, 12 weeks, 24 weeks
  Accommodation facility measured with accommodative flipper
Changes in accommodation function | 1 weeks, 4weeks, 12 weeks, 24 weeks
  Accommodation function including accommodation amplitude, accommodation response, positive relarive accommodation, and negative relative accommodation measured with phoropter
Change in accommodation convergence to accommodation(AC/A) ratio | 1 weeks, 4weeks, 12 weeks, 24 weeks
  AC/A ratio measured with synoptophore

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
We concerns about patient privacy issues and it's better to protect the publication potential.